CLINICAL TRIAL: NCT01593618
Title: Empowering Cancer Survivors Through Information Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007NT078
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Cancer Survivor
Keywords: cancer survivor
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-Based Intervention (Experimental): UMFollowUp - web-based internet resource for information about their diagnostic histories, recommendations for follow-up care, and tips to enhance their treatment, psychosocial and physical well-being.
  Interventions: Behavioral: UMFollowUp
- Standard of Care (Active Comparator): Patients will receive information regarding their diagnosis, treatments, and ongoing health needs from their provider, but will not be provided access to the website.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: UMFollowUp — Web-based internet resource for self-reported treatment summaries and psychosocial and physical well-being.
  Arms: Web-Based Intervention
Other: Standard of Care — Patients will receive information regarding their diagnosis, treatments, and ongoing health needs from their provider, but will not be provided access to the website.
  Arms: Standard of Care

SUMMARY:
This is a randomized controlled trial of a web-based informational intervention (UMFollowUp) for adolescent and young adult survivors of childhood cancer to improve cancer knowledge and psychosocial functioning.

DETAILED DESCRIPTION:
Individuals randomly assigned to the control group will receive standard of care for the duration of their participation. This means they will continue to receive information regarding their diagnosis, treatments and ongoing health needs from their provider (no access to website).

Individuals randomly assigned to the treatment group will receive access to UMFollowUp, a secure, HIPAA-compliant website.

All participants will be asked to complete paper-and-pencil surveys at baseline and 9 months later to determine the impact of the web-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* History of diagnosis of hematologic malignancy or malignant neoplasm, and in disease free remission at time of recruitment.
* Must be English-speaking and have access to a computer with internet access, and must have completed treatment at University of Minnesota Medical Center-Fairview for cancer.

Exclusion Criteria:

* Individual with significant visual impairments and neurologic/cognitive difficulties which limit their ability to see and under our outcome questionnaires or website content will be excluded from participation.

Ages: 15 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2007-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Cancer Knowledge Survey | Time of Enrollment and 9 Months Later
  Measure of patient reported knowledge of their cancer diagnosis, history and treatments.

SECONDARY OUTCOMES:
SF-36 Questionnaire | Time of Enrollment and 9 Months Later
  A measure of quality of life.
Cancer Rehabilitation Evaluation System | Time of Enrollment and 9 Months Later
  Short Form (SF) Medical Interaction Subscale
Herth Hope Index | Time of Enrollment and 9 Months Later
  A measure of self-reported hope.
Multidimensional Scale of Perceived Social Support | Time of Enrollment and 9 Months Later
  A measure of self-reported social support.
Health Locus of Control Scale | Time of Enrollment and 9 Months Later
  A measure of self-reported locus of control.
State Trait Anxiety Inventory | Time of Enrollment and 9 Months Later
  A measure of self-reported anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Kunin-Batson, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States